CLINICAL TRIAL: NCT04575272
Title: Ultrasound-guided Deep Versus Superficial Continuous Serratus Anterior Plane Block for Pain Management in Patients With Multiple Rib Fractures: Randomized Double-blind Clinical Trial
Brief Title: Ultrasound-guided Deep Versus Superficial Continuous Serratus Anterior Plane Block for Pain Management in Patients With Multiple Rib Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed mamdouh mohammed mahmoud, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Serratus Plane Block and MFRs
Record Dates: First submitted 2020-09-20; First posted 2020-10-05 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Multiple Rib Fractures; Pain, Acute; Serratus Anterior Plane Block
Keywords: serratus anterior plane block; multiple rib fractures
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: neither the patient or the investigator included in data collection will be aware of the type of block performed or the group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Deep Serratus Anterior Plane Block group (Experimental): at the level of the fifth rib in the mid-axillary line. After anaesthetizing the skin with 2 mL of lidocaine 2%, an 18-gauge Touhy needle was introduced in-plane, under direct visualization, to the plane immediately deep to the serratus anterior muscle. After negative aspiration, 35 mL of bupivacaine 0.25% will be injected. Afterwards, a 20-gauge peripheral nerve catheter will be threaded into the space. then bupivacaine 0.125% infusion at a rate of 5 ml/h by an Infusion Syringe Pump will be started.
  Interventions: Procedure: Ultrasound-guided continuous serratus anterior plane block
- Continuous Superficial Serratus Anterior Plane Block group (Active Comparator): at the level of the fifth rib in the mid-axillary line. After anaesthetizing the skin with 2 mL of lidocaine 2%, an 18-gauge Touhy needle was introduced in-plane, under direct visualization, to the plane immediately superficial to the serratus anterior muscle. After negative aspiration, 35 mL of bupivacaine 0.25% will be injected. Afterwards, a 20-gauge peripheral nerve catheter will be threaded into the space. then bupivacaine 0.125% infusion at a rate of 5 ml/h by an Infusion Syringe Pump will be started.
  Interventions: Procedure: Ultrasound-guided continuous serratus anterior plane block

INTERVENTIONS:
Procedure: Ultrasound-guided continuous serratus anterior plane block — Local anesthetic infusion though a peripheral nerve catheter placed related to the serratus anterior muscle at the level of the 5th rib

SUMMARY:
The present clinical study will be undertaken to evaluate the effect of Ultrasound-guided Deep versus Superficial continuous Serratus Anterior Plane Block for pain management in patients with multiple rib fractures.

DETAILED DESCRIPTION:
Thoracic blunt trauma, especially when multiple rib fractures are associated, is challenging to manage and causes significant morbidity due to the severe pain implied.

Patients can present with respiratory compromise as their capacity to expand the thorax is limited by pain. As a result, they are at high risk to develop atelectasis and pneumonia.

the key goal of management is adequate analgesia and pulmonary volume expansion Various strategies to treat such pain have been utilized, including regional analgesia (intrapleural, intercostal paravertebral nerve blockade), and neuraxial analgesia (thoracic epidural analgesia (TEA), intrathecal opioids).

The use of neuraxial analgesia in polytrauma is frequently limited by the need for aggressive venous thromboembolic (VTE) prophylaxis, and positioning of the patient for a neuraxial approach may be impossible.

There is a growing interest in exploring treatments that are less invasive than EA and can be performed on patients who have contraindications to neuraxial analgesia. Ultrasound-guided Serratus Anterior Plane (SAP) block is a recent technique, first described by Blanco et al. in 2013, that provides analgesia for the thoracic wall by blocking the lateral branches of the intercostal nerves from T2 to L2. It is a safe, simple to perform block with no significant contraindications or side effects. he described 2 potential spaces, one superficial and another deep to serratus. The SAPB has been used effectively for the management of pain in the context of rib fractures, thoracoscopic surgery, thoracotomy, breast surgery, and post-mastectomy pain syndrome, few studies compared the two approaches, and the difference between them has not yet been studied in patients with multiple rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex, having three or more unilateral fracture ribs and admitted to the trauma ICU, Rib fractures were confirmed by X-ray and CT scan reads.

Exclusion Criteria:

* significant head injury and unconsciousness (GCS less than 14)
* Patients with significant pain from other injuries
* pathological obesity (body mass index ≥35)
* history of drug allergy local anesthetics
* local infection at the injection site
* inability to obtain consent from patient or surrogate, and patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Change in pain score | before and after the block at "30 minutes", "2hours", "4hours", "6hours", "12hours", "24hours", "36hours", "48 hours" & "72hours"
  patient report numerical rating scale (NRS) 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable"

SECONDARY OUTCOMES:
Change in inspiratory volumes (mL) | before and after block at "90 minutes" then every "12hours" for 3 days
  Maximum inspiratory respiratory volume (measured in ml) recorded on single use of incentive spirometer device
change in Serum beta-endorphin level | before procedure and at 24 hours post procedure
  We will use radioimmunoassays to measure plasma beta-endorphin level
Lung Ultrasound Score (LUSS) | before and after block at "90 minutes" then every "24 hours" for 3 days
  We will use a techniques based on the international evidence-based recommendations for point-of-care lung ultrasound that recommended using a complete eight-zone lung ultrasound ,The worst ultrasound pattern observed in each zone was recorded and used to calculate the sum of the scores (total score = 24).
mean arterial blood pressure | before and after the block every "2hours" for 3 days
  mean arterial blood pressure by non invaisive blood pressure monitoring
heart rate | before and after the block every "2hours" for 3 days
  heart rate by EKG monitor
peripheral arterial oxygen saturation (SpO2) | before and after the block every "2hours" for 3 days
  measured by Pulse oximetry

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] May L, Hillermann C, Patil S. Rib fracture management. BJA Educ. 2016 Jan 1;16(1):26-32.
- [Background] Chien CY, Chen YH, Han ST, Blaney GN, Huang TS, Chen KF. The number of displaced rib fractures is more predictive for complications in chest trauma patients. Scand J Trauma Resusc Emerg Med. 2017 Feb 28;25(1):19. doi: 10.1186/s13049-017-0368-y. PMID 28241883
- [Background] Lotfipour S, Kaku SK, Vaca FE, Patel C, Anderson CL, Ahmed SS, Menchine MD. Factors associated with complications in older adults with isolated blunt chest trauma. West J Emerg Med. 2009 May;10(2):79-84. PMID 19561823
- [Background] Vasigh A, Jaafarpour M, Khajavikhan J, Khani A. The Effect of Gabapentin Plus Celecoxib on Pain and Associated Complications After Laminectomy. J Clin Diagn Res. 2016 Mar;10(3):UC04-8. doi: 10.7860/JCDR/2016/17923.7346. Epub 2016 Mar 1. PMID 27134973
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192
- [Background] Hernandez N, de Haan J, Clendeninn D, Meyer DE, Ghebremichael S, Artime C, Williams G, Eltzschig H, Sen S. Impact of serratus plane block on pain scores and incentive spirometry volumes after chest trauma. Local Reg Anesth. 2019 Aug 2;12:59-66. doi: 10.2147/LRA.S207791. eCollection 2019. PMID 31447581
- [Background] Okmen K, Okmen BM. The efficacy of serratus anterior plane block in analgesia for thoracotomy: a retrospective study. J Anesth. 2017 Aug;31(4):579-585. doi: 10.1007/s00540-017-2364-9. Epub 2017 Apr 26. PMID 28447227
- [Background] Beard L, Hillermann C, Beard E, Millerchip S, Sachdeva R, Gao Smith F, Veenith T. Multicenter longitudinal cross-sectional study comparing effectiveness of serratus anterior plane, paravertebral and thoracic epidural for the analgesia of multiple rib fractures. Reg Anesth Pain Med. 2020 May;45(5):351-356. doi: 10.1136/rapm-2019-101119. Epub 2020 Mar 11. PMID 32165553
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Durant E, Dixon B, Luftig J, Mantuani D, Herring A. Ultrasound-guided serratus plane block for ED rib fracture pain control. Am J Emerg Med. 2017 Jan;35(1):197.e3-197.e6. doi: 10.1016/j.ajem.2016.07.021. Epub 2016 Jul 19. No abstract available. PMID 27595172
- [Background] Piracha MM, Thorp SL, Puttanniah V, Gulati A. "A Tale of Two Planes": Deep Versus Superficial Serratus Plane Block for Postmastectomy Pain Syndrome. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):259-262. doi: 10.1097/AAP.0000000000000555. PMID 28079733
- [Background] Zocca JA, Chen GH, Puttanniah VG, Hung JC, Gulati A. Ultrasound-Guided Serratus Plane Block for Treatment of Postmastectomy Pain Syndromes in Breast Cancer Patients: A Case Series. Pain Pract. 2017 Jan;17(1):141-146. doi: 10.1111/papr.12482. Epub 2016 Sep 2. PMID 27587333
- [Background] Bhoi D, Selvam V, Yadav P, Talawar P. Comparison of two different techniques of serratus anterior plane block: A clinical experience. J Anaesthesiol Clin Pharmacol. 2018 Apr-Jun;34(2):251-253. doi: 10.4103/joacp.JOACP_294_16. No abstract available. PMID 30104841
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031